CLINICAL TRIAL: NCT07220083
Title: A Multicentre, Randomised, Double-blind, Parallel Group, Placebo-controlled Trial to Assess the Effects of Oral TRPC6 Inhibitor BI 764198 Taken Over a 104 Week Treatment Period in Adult and Adolescent Participants With Primary Focal Segmental Glomerulosclerosis (pFSGS) or Genetic FSGS Related to TRPC6 Gene Variants
Brief Title: A Study to Find Out if BI 764198 Helps Adults and Adolescents With a Kidney Condition Called Focal Segmental Glomerulosclerosis (FSGS)
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1434-0017; 2025-522191-86 (Registry Identifier: CTIS (EU)); U1111-1326-1647 (Registry Identifier: WHO International Clinical Trials Registry Platform (ICTRP))
Record Dates: First submitted 2025-10-22; First posted 2025-10-23 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Focal Segmental Glomerulosclerosis
MeSH Terms: conditions — Glomerulosclerosis, Focal Segmental

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BI 764198 treatment (Experimental)
  Interventions: Drug: BI 764198
- Placebo treatment (Experimental)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BI 764198 — BI 764198
  Arms: BI 764198 treatment
Drug: Placebo — Placebo matching BI 764198
  Arms: Placebo treatment

SUMMARY:
This study is open to adults and adolescents with a kidney condition called focal segmental glomerulosclerosis (FSGS). The purpose of this study is to find out whether a medicine called BI 764198 helps people with FSGS.

Participants are put into 2 groups randomly, which means by chance. Every participant has an equal chance of being in each group. One group takes BI 764198 tablets, and the other group takes placebo tablets. Placebo tablets look like BI 764198 tablets but do not contain any medicine.

Participants take a tablet once a day for up to 2 years. All participants also continue their standard medication for FSGS.

Participants are in the study for up to 2 years. During this time, they visit the study site about every 3 months. Participants regularly collect urine samples. This is done to check their kidneys. The results are compared between the two groups to see whether the treatment works. The doctors also regularly check participants' health and take note of any unwanted effects.

ELIGIBILITY:
Inclusion criteria:

1. Male or female participants ≥12 years old on the day of signing informed consent/assent (Visit 1)
2. Weight of ≥40 kg at the screening visit (Visit 1)
3. Body mass index (BMI) of ≤40 kg/m² at the screening visit (Visit 1)
4. Participants with a diagnosis prior to the screening visit (Visit 1) of either:

   * Biopsy-confirmed primary focal segmental glomerulosclerosis (pFSGS) (based on Investigator's judgement) OR
   * Genetic focal segmental glomerulosclerosis (FSGS) resulting from a gain-of-function mutation in the transient receptor potential cation subfamily C member 6 (TRPC6) gene (based on historical genetic test)
5. Urine protein-creatinine ratio (UPCR) ≥1500 mg/g based on the mean of the spot urine sample and first morning void urine sample (both assessed by central laboratory) at the screening visit (Visit 1)
6. Estimated glomerular filtration rate (eGFR)

   * For adult participants (≥18 years): ≥25 mL/min/1.73 m² (chronic kidney disease epidemiology collaboration (CKD-EPI) formula based on combined serum creatinine plus cystatin C) at the screening visit (Visit 1)
   * For adolescent participants (12 to <18 years); ≥25 mL/min/1.73 m² based on chronic kidney disease under 25 years (CKiD U25) formula using height and serum cystatin C at the screening visit (Visit 1) Further inclusion criteria apply.

Exclusion criteria:

1. Known monogenic or syndromic causes of FSGS (with the exception of TRPC6 gain-of-function gene mutations)
2. Clinical or histologic evidence of secondary maladaptive or toxic forms of FSGS (based on Investigator's judgement)
3. FSGS of undetermined cause (FSGS-UC) with a diagnosis prior to the screening visit (Visit 1) (based on Investigator's judgement)
4. A history of organ transplantation or planned organ transplantation during the course of the trial
5. Use of intravenous immunosuppressive agents (e.g. cyclophosphamide, rituximab, obinutuzumab) in the last 6 months prior to screening (Visit 1) Further exclusion criteria apply.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 286 (Estimated)
Dates: Start 2026-02-06 (Estimated); Primary Completion 2029-11-20 (Estimated); Study Completion 2029-12-18 (Estimated)

PRIMARY OUTCOMES:
Relative change in 24-hour urinary protein-to-creatinine ratio (UPCR, measured in mg/g) from baseline to Week 104 | Baseline and Week 104

SECONDARY OUTCOMES:
Key secondary endpoint: Absolute change in eGFRcys in mL/min/1.73m2 from baseline to Week 104 | Baseline and Week 104
  Estimated glomerular filtration rate based on serum cystatin C (eGFRcys)
Key secondary endpoint: Treatment response, defined as 24-hr UPCR <1000 mg/g at Week 104 | At Week 104
  24-hour urinary protein-to-creatinine ratio (24-hr UPCR)
Treatment response, defined as 24-hr UPCR <1000 mg/g and eGFRcys ≥85% vs. baseline at Week 104 and no treatment failure between randomisation and Week 104 (combined or multi-component endpoint) | At Week 104
  24-hour urinary protein-to-creatinine ratio (24-hr UPCR), Estimated glomerular filtration rate based on serum cystatin C (eGFRcys).
  Treatment failure defined as one or more of the following:
  * Use of rescue therapy due to worsening or severely active disease leading to the Investigator concluding that the randomised treatment regimen has failed and requires additional treatment.
  * Presence of any of the following events:
    * End-stage renal disease
    * Receipt of a kidney transplant
    * Death
  * Intensification of concomitant medication used at screening. Therapies that are considered include:
    * Calcineurin inhibitors
    * Azathioprine
    * Mycophenolate mofetil
    * Glucocorticoids: Prednisolone dose escalated to a dose of ≥20 mg/d (oral or intravenous) or equivalent for more than 14 days for treatment of kidney disease
Complete remission, defined as 24-hr UPCR <300 mg/g at Week 104 | At Week 104
  24-hour urinary protein-to-creatinine ratio (24-hr UPCR)
Change from baseline across disease-specific clinical outcome assessment (COA) NS-SIM-PRO at Week 104 | Baseline and Week 104
  The nephrotic syndrome swelling impact measure (NS-SIM-PRO) has 23 items covering physical function (e.g. mobility), physical symptoms (e.g. fatigue, nausea), and essential function (e.g. vision) impacts identified as being important aspects of participants' experiences with nephrotic-syndrome related swelling.
  It is expected that all item responses will be combined to generate a single score representing overall swelling impact.
  The score ranges from 0 up to 4 (0 = never, 1 = almost never, 2 = sometimes, 3 = often, 4 = almost always). A lower score on any of the NS-SIM-PRO subscales indicate a better quality of life.
  The NS-SIM-PRO is applicable only for participants where the investigator confirms the participant is suffering from the symptom swelling at the time of assessment.
Change from baseline across clinical outcome assessment (COA) KDQOL-36 at Week 104 | Baseline and Week 104
  Kidney disease quality of life 36-item short form survey (KDQOL-36) assessing the health-related quality of life (HRQOL) in adult participants with kidney disease. It combines the generic SF-12 Health Survey with additional items specifically relevant to kidney disease.
  Key Components:
  * SF-12 Health Survey: Includes 12 items that measure physical and mental health, providing a broad overview of the patient's general health status.
  * Burden of Kidney Disease: This subscale (4 items) assesses how much kidney disease interferes with daily life and causes frustration.
  * Symptoms/Problems: This subscale (12 items) evaluates the frequency and severity of symptoms related to kidney disease, such as pain, fatigue, and sleep disturbances.
  * Effects of Kidney Disease: This subscale (8 items) measures the impact of kidney disease on daily activities and overall well-being.
  The score ranges from 0 up to 6 and a higher score on most of the KDQOL-36 subscales indicate a better quality of life.

CONTACTS AND LOCATIONS:
Locations (205):
- United States (40):
  - Alabama Kidney Research, Alabaster, Alabama
  - Nephrology Consultants, LLC, Huntsville, Alabama
  - Southwest Kidney Institute, Surprise, Arizona
  - Amicis Research Center - Balboa, Granada Hills, California
  - Academic Medical Research Institute - Glendale, Los Angeles, California
  - North America Research Institute, San Dimas, California
  - Kaiser Permanente - French Campus, San Francisco, California
  - Valiance Clinical Research-Tarzana-68237, Tarzana, California
  - National Institute of Clinical Research - Victorville, Victorville, California
  - Colorado Kidney Center, Denver, Colorado
  - Total Research Group, LLC, Miami, Florida
  - CTR Oakwater, LLC, Orlando, Florida
  - Panoramic Health, Riverview, Florida
  - Emory Children's Center, Atlanta, Georgia
  - Memorial Health University Hospital, Savannah, Georgia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Endeavor Health, Evanston, Illinois
  - Wichita Nephrology Group, Wichita, Kansas
  - Northwest Louisiana Nephrology, Shreveport, Louisiana
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Henry Ford Hospital, Detroit, Michigan
  - Elixia MKC, LLC, Pontiac, Michigan
  - St. Clair Nephrology Research, LLC - Shelby Township, Utica, Michigan
  - Mayo Clinic, Rochester, Rochester, Minnesota
  - Elixia MNA, LLC, City of Saint Peters, Missouri
  - DaVita Clinical Research-Las Vegas-67781, Las Vegas, Nevada
  - New York Nephrology and Dialysis Access Surgery, PC, Clifton Park, New York
  - NYU Langone Nephrology Associates-Mineola, Mineola, New York
  - Duke University Medical Center, Durham, North Carolina
  - Brookview Hills Research Associates LLC, Winston-Salem, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Northeast Clinical Research Center, Bethlehem, Pennsylvania
  - Clinical Renal Associates, Exton, Pennsylvania
  - Southeast Renal Research Institute, Chattanooga, Tennessee
  - Texas Tech University Health Sciences Center-Amarillo-63885, Amarillo, Texas
  - Nephrotex Research Group, Dallas, Texas
  - Provecta Researh Network, Houston, Texas
  - Utah Kidney Research Institute, Salt Lake City, Utah
  - Virginia Nephrology, Arlington, Virginia
  - West Virginia University Medicine, Morgantown, West Virginia
- Argentina (7):
  - Terapia Renal Domiciliaria, Buenos Aires
  - Hospital Italiano de Buenos Aires, CABA
  - CEMIC, CABA
  - Centro Medico Dra Laura Maffei, Ciudad Autonoma Buenos Aires
  - Clinica Privada Velez Sarfield, Córdoba
  - Hospital Universitario Austral, Pilar
  - CardioAlem Investigaciones, San Isidro
- Australia (4):
  - Nepean Hospital, Kingswood, New South Wales
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Griffith Health, Southport, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
- Belgium (3):
  - AZORG Ziekenhuis, Aalst
  - UZ Leuven, Leuven
  - Centre Hospitalier Universitaire de Liège, Liège
- Brazil (6):
  - Synvia, Campinas
  - Universidade Federal do Ceará, Fortaleza
  - Hospital de Clínicas de Porto Alegre, Porto Alegre
  - Hospital das Clínicas da Universidade Federal de Pernambuco, Recife
  - Fundação Oswaldo Ramos (Hospital do Rim), São Paulo
  - Centro de Pesquisa Clínica de Nefrologia do ICHC, São Paulo
- Canada (2):
  - Victoria Hospital (LHSC), London, Ontario
  - Maisonneuve-Rosemont Hospital, Montreal, Quebec
- China (21):
  - The First Affiliated Hospital of Baotou Medical College, Baotou
  - Peking University First Hospital, Beijing
  - Beijing Tsinghua Changgung Hospital, Beijing
  - The Second Hospital of Jilin University, Changchun
  - The Second Xiangya Hospital Of Central South University, Changsha
  - West China Hospital, Sichuan University, Chengdu
  - People's Hospital of Sichuan Province, Chengdu
  - Guangdong Provincial People's Hospital, Guangzhou
  - Guizhou People's Hospital, Guiyang
  - The First Affiliated Hospital, Zhejiang University, Hangzhou
  - Lanzhou University Second Hospital, Lanzhou
  - The First Affiliated Hospital of Nanchang University, Nanchang
  - Zhongda Hospital Southeast University, Nanjing
  - The First People's Hospital of Nanning, Nanning
  - The First Affiliated Hospital of Guangxi Medical University, Nanning
  - Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai
  - Shanghai General Hospital, Shanghai
  - Shanxi Provincial People's Hospital, Taiyuan
  - Renmin Hospital of Wuhan University, Wuhan
  - First Affiliated Hospital of Xi'an JiaoTong University, Xi'an
  - Zhongshan Hospital Affiliated to Xiamen University, Xiamen
- Croatia (2):
  - Clinical Hospital Sveti Duh, Zagreb
  - Poliklinika Bonifarm Zagreb, Zagreb
- Denmark (2):
  - Copenhagen University Hospital, Rigshospitalet, København Ø
  - Zealand University Hospita; Roskilde, Roskilde
- France (9):
  - CHU Amiens-Picardie, Amiens
  - HOP Pellegrin, Bordeaux
  - HOP de la Cavale Blanche, Brest
  - Hôpital Henri Mondor, Créteil
  - HOP Edouard Herriot, Lyon
  - HOP Pasteur, Nice
  - HOP Nîmes, Nîmes
  - Hôpital Necker, Paris
  - HOP Nancy, Vandœuvre-lès-Nancy
- Germany (7):
  - Vivantes Klinikum im Friedrichshain, Berlin
  - Universitätsklinikum Köln (AöR), Cologne
  - Universitätsklinikum Hamburg, Eppendorf, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Universitätsklinikum Heidelberg, Heidelberg
  - Universität Leipzig, Leipzig
  - Universitätsmedizin der Johannes Gutenberg-Universität Mainz, Mainz
- Greece (2):
  - University General Hospital of Heraklion, Heraklion
  - Univ. Gen. Hosp. of Patras, Pátrai
- Queen Mary Hospital, Hong Kong, Hong Kong
- India (4):
  - Aartham Multi Super Speciality Hospital, Ahmedabad
  - AIIMS Bhubaneshwar, Bhubaneshwar
  - Government Medical College, Kozhikode
  - Noble Hospital Pvt Ltd, Pune
- Italy (6):
  - Azienda Universitaria Ospedaliera Consorziale Policlinico Bari, Bari
  - Policlinico S. Orsola-Malpighi, Bologna
  - Asst Santi Paolo E Carlo, Milan
  - Azienda Ospedaliera Universitaria Policlinico Paolo Giaccone, Palermo
  - Fondazione Salvatore Maugeri, Pavia
  - ASST dei Sette Laghi, Varese
- Japan (14):
  - Kasugai Municipal Hospital, Aichi, Kasugai
  - Daido Clinic, Aichi, Nagoya
  - Japanese Red Cross Aichi Medical Center Nagoya Daini Hospital, Aichi, Nagoya
  - Chiba University Hospital, Chiba, Chiba
  - National Hospital Organization Chibahigashi National Hospital, Chiba, Chiba
  - Japanese Red Cross Fukuoka Hospital, Fukuoka, Fukuoka
  - Kurume University Hospital, Fukuoka, Kurume
  - Kobe University Hospital, Hyogo, Kobe
  - Saiseikai Yokohamashi Nanbu Hospital, Kanagawa, Yokohama
  - Nara Prefecture General Medical Center, Nara, Nara
  - Dokkyo Medical University Saitama Medical Center, Saitama, Koshigaya
  - Institute of Science Tokyo Hospital, Tokyo, Bunkyo-ku
  - The Jikei University Hospital, Tokyo, Minato-ku
  - Tokyo Women's Medical University Hospital, Tokyo, Shinjuku-ku
- Malaysia (3):
  - Hospital Kuala Lumpur, Kuala Lumpur
  - University of Malaya Medical Centre, Lembah Pantai
  - Sunway Medical Centre, Subang Jaya
- Mexico (6):
  - Centenario Hospital Miguel Hidalgo, Aguascalientes
  - Health Pharma Professional Research S.A. de C.V., Mexico City
  - Soltmed Smo, Mexico City
  - Instituto Nacional de Cardiologia Ignacio Chavez, Mexico City
  - Instituto Nacional de Cs Médicas y Nutrición S Zubiran, Mexico City
  - Servicios de Oncología Médica Integral, S.A. de C.V. Sucursal Renal, Monterrey
- Netherlands (3):
  - Amsterdam UMC Locatie AMC, Amsterdam
  - Universitair Medisch Centrum Groningen, Groningen
  - Radboud Universitair Medisch Centrum, Nijmegen
- New Zealand (2):
  - Optimal Clinical Trials - Christchurch, Christchurch
  - Optimal Clinical Trials North, Rosedale, Auckland
- Norway (4):
  - Akershus Universitetssykehus HF, Lørenskog
  - Oslo Universitetssykehus HF, Ullevål sykehus, Oslo
  - Helse Stavanger, Stavanger Universitetssykehus, Stavanger
  - Universitetssykehuset Nord-Norge, Tromsø, Tromsø
- Poland (4):
  - Centralny Szpital Kliniczny Uniwersytetu Medycznego w Łodzi, Lodz
  - Uniwersytet Medyczny im. Karola Marcinkowskiego w Poznaniu, Poznan
  - Pomorski Uniwersytet Medyczny w Szczecinie, Samodzielny Publiczny Szpital Kliniczny nr 2, Szczecin
  - Centralny Szpital Kliniczny MON WIM, Warsaw
- Portugal (10):
  - ULS de Almada -Seixal, E. P. E. - Hospital Garcia de Orta, Almada
  - ULS de Amadora/ Sintra, E.P.E. - Hospital Professor Doutor Fernando Fonseca, Amadora
  - ULS Braga, Braga
  - CHUC - Centro Hospitalar e Universitário de Coimbra, EPE, Coimbra
  - ULS de São José, Lisbon
  - ULS de Santa Maria, E.P.E, Lisbon
  - Unidade Local de Saúde Lisboa Occidental, E.P.E, Lisbon
  - ULS de Loures-Odivelas, E.P.E, Loures
  - ULS de Santo Antônio, E.P.E - Centro Hospitalar Universitário de Santo António, Porto
  - Unidade Local de Saúde da Arrábida,E.P.E, Setúbal
- Romania (2):
  - Institutul Clinic Fundeni, Bucharest
  - Cluj Napoca Clinical County Hospital, Cluj-Napoca
- Singapore (3):
  - National University Hospital, Singapore
  - Singapore General Hospital, Singapore
  - Tan Tock Seng Hospital, Singapore
- Slovakia (2):
  - Univerzitna nemocnica L. Pasteura Kosice, Košice
  - Univ. Hospital Martin, Martin
- South Korea (5):
  - Pusan National University Hospital, Busan
  - Samsung Medical Center, Gangnam-gu
  - Inje University Ilsan Paik Hospital, Goyang
  - Severance Hospital, Seoul
  - Ajou University Hospital, Suwon
- Spain (8):
  - Complejo Hospitalario Torrecárdenas, Almería
  - Hospital del Mar, Barcelona
  - Hospital Universitari Vall D Hebron, Barcelona
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital Sant Joan de Déu, Barcelona
  - Hospital Universitario Virgen de las Nieves, Granada
  - Hospital Clínico San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
- Sweden (5):
  - Danderyds Sjukhus, Danderyd
  - Universitetssjukhuset, Linköping, Linköping
  - Skånes universitetssjukhus, Lund
  - Karolinska Universitetssjukhuset, Stockholm
  - Uppsala University Hospital, Uppsala
- University Hospital Bern, Bern, Switzerland
- Taiwan (6):
  - Buddhist Tzu Chi General Hospital-Hualien-20741, Hualien City
  - Taipei Medical University-Shuang Ho Hospital, New Taipei City
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
- Turkey (Türkiye) (6):
  - Adana City Hospital, Adana
  - Ankara Etlik City Hospital, Ankara
  - Bursa Uludag University, Bursa
  - İstanbul Çapa University, Istanbul
  - Kocaeli University Faculty of Medicine Hospital, İzmit
  - Erciyes University, Melikgazi/Kayseri
- United Kingdom (5):
  - Clatterbridge Hospital, Bebington
  - Bradford Institute for Health Research, Bradford
  - Leicester General Hospital, Leicester
  - King's College Hospital, London
  - Salford Royal, Salford

IPD SHARING:
Plan to Share IPD: Yes
Once the criteria in section 'time frame' are fulfilled, researchers can use the following link https://www.clinicalstudies.boehringer-ingelheim.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement". Furthermore, researchers can request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: One year after the approval has been granted by major Regulatory Authorities and after the primary manuscript has been accepted for publication, or after termination of the development program.
Access Criteria: For study documents -upon signing of a 'Document Sharing Agreement'.For study data -1. after the submission and approval of the research proposal (checks will be performed by the sponsor and/or the independent review panel, including checking that the planned analysis does not compete with sponsor'spublication plan); 2. and upon signing of a legal agreement.
URL: https://www.clinicalstudies.boehringer-ingelheim.com/msw/datasharing

REFERENCES:
- See also: Related Info — https://www.clinicalstudies.boehringer-ingelheim.com/msw/datatransparency